CLINICAL TRIAL: NCT06477237
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of HB0017 Injection in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Study of Efficacy and Safety of HB0017 in Patients With Moderate to Severe Plaque Psoriasis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HB0017-07
Record Dates: First submitted 2024-06-18; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Psoriasis
Keywords: psoriasis; HB0017
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HB0017 (Experimental): Participants will receive HB0017 at week 0,1,2,4,8 followed by once every four weeks (Q4W) or once every eight weeks (Q8W) at Week 12.
  Interventions: Biological: HB0017 Q4W; Biological: HB0017 Q8W
- placebo (Placebo Comparator): Participants will receive placebo at week 0,1,2,4,8 followed by HB0017 once every four weeks (Q4W) at Week 12.
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: HB0017 Q4W — HB0017 at W0,1,2,4,8+HB0017Q4W
  Arms: HB0017
Biological: HB0017 Q8W — HB0017 at W0,1,2,4,8+HB0017Q8W
  Arms: HB0017
Biological: placebo — placebo at W0,1,2,4,8+HB0017Q4W
  Arms: placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, phase III clinical study which is designed to determine the efficacy, safety, immunogenicity and pharmacokinetics, and pharmacodynamics of HB0017 Injection in the treatment of moderate to severe plaque psoriasis in adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-75 years (inclusive)
* Chronic plaque psoriasis (PSO) for at least 6 months prior to the Randomization.
* Psoriasis Area Severity Index (PASI) >=12 and body surface area (BSA) affected by PSO >=10% and Static Physician Global Assessment (sPGA) score >=3.
* Subjects who are suitable for systemic treatment or phototherapy for psoriasis as judged by the investigator
* Subjects who are able to use effective contraception from the screening period to 6 months after the last dose

Key Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and/or guttate psoriasis) at screening or baseline
* Drug-induced psoriasis
* Ongoing use of prohibited treatments
* Any active infection (other than common cold) within 14 days
* Serious infection defined as requiring hospitalization or iv anti-infective(s) within 1 month prior to randomization
* Have previously received any drug that directly targets IL-17 or IL-17 receptor
* Have concurrent or recent use of any biologic agent within the following washout periods: etanercept <28 days; infliximab and adalimumab <60 days; golimumab < 90 days; anti-IL-12/anti-IL-23 or anti-IL-23p19 antibody drugs <6 months; or other anti-psoriatic therapy not listed herein within its 5 half-lives prior to randomization
* A history of inflammatory bowel disease or other serious autoimmune disease
* Previously diagnosed with serious mental illness such as anxiety, depression or suicidal tendency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving PASI 75 response at Week 12 | Week 12
  The PASI75 response assessments are based on at least 75% improvement in PASI score from Baseline.
Proportion of subjects achieving sPGA 0/1 response at Week 12 | Week 12
  The sPGA is a physician's determination of the participant's psoriasis lesions overall at a given time point categorized by descriptions for induration, erythema, and scaling. For the analysis of responses, the participant's psoriasis is assessed as clear (0), Almost clear (1), mild (2), moderate (3), severe (4). An sPGA 0/1 response was defined as a post-baseline sPGA score of 0 or 1.

SECONDARY OUTCOMES:
Proportion of subjects achieving PASI 90 response at Week 12 | Week 12
  The PASI90 response assessments are based on at least 90% improvement in PASI score from Baseline.
PASI 90 response maintainance at week 52 | Week12-52
  Proportion of subjects maintaining PASI 90 response at Week 52 among those with PASI 90 response at Week 12
sPGA 0/1 response maintainance at week 52 | Week 12-52
  Proportion of subjects maintaining sPGA 0/1 response at Week 52 among those with sPGA 0/1 response at Week 12.
PASI 75 response maintainance at week 52 | Week12-52
  Proportion of subjects maintaining PASI 75 response at Week 52 among those with PASI 75 response at Week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, MD, Principal Investigator — Peking University People's Hospital
Locations (44):
- China (44):
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Nanyang First People's Hospital, Nanyang, Henan
  - Beijing Friendship Hospital, Beijing
  - China-Japan Friendship hospital, Beijing
  - Peking University People's Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Jilin University Second Hospital, Changchun
  - The first hospital of Jilin University, Changchun
  - Xiangya Hospital of Central South University, Changsha
  - Affiliated Hospital of Chengde Medical University, Chengde
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital of Sichuan University, Chengdu
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing
  - Dongguan People's Hospital, Dongguan
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Dermatology Hospital of Southern Medical University, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - Hangzhou Third People's Hospital, Hangzhou
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - Jiaxing First Hospital, Jiaxing
  - Shandong Dermatology Hospital, Jinan
  - Jining First People's Hospital, Jining
  - The First Affiliated Hospital of Kunming Medical University, Kunming
  - The Second Affiliated Hospital of Kunming Medical University, Kunming
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Dermatology Hospital of Jiangxi Province, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu University Affiliated Hospital, Nanjing
  - Ningbo Second Hospital, Ningbo
  - Shanghai Dermatology Hospital, Shanghai
  - People's Hospital of Liaoning Province, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - Shiyan People's Hospital, Shiyan
  - The Second Hospital of Shanxi Medical University, Taiyuan
  - Wenzhou Medical University Affiliated First Hospital, Wenzhou
  - Wuhan University People's Hospital, Wuhan
  - The First Affiliated Hospital of Wannan Medical College, Wuhu
  - Wuxi Second People's Hospital, Wuxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xingtai People's Hospital, Xingtai
  - Yangjiang People's Hospital, Yangjiang